CLINICAL TRIAL: NCT07196930
Title: Valvular Heart Disease in Women Registry
Acronym: VHD-W
Status: Recruiting | Type: Observational
Sponsor: Valvular Heart Disease in Women Registry (Network)
Collaborators: European Association of Cardiovascular Imaging (Other)
Responsible Party: Principal Investigator, Julia Grapsa, Professor, Cardiovascular Medicine, Valvular Heart Disease in Women Registry
Other Study IDs: VHD-W Registry
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Valve Disease, Heart; Gender Bias; Guideline Adherence; Guideline Implementation; Disparities; Registry
Keywords: valvular heart disease; registry; cardiovascular disease; gender disparities; Guidelines adherence
MeSH Terms: conditions — Heart Valve Diseases; Sexism; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with Valvular Heart Disease: Women with Valvular Heart Disease
- Men with Valvular Heart Disease: Men with Valvular Heart Disease

SUMMARY:
Valvular heart disease (VHD) is a major global health issue. Untreated rheumatic heart disease persists in many regions, preventable with timely care. Higher-income countries face rising calcific valve disease from aging, worsened by VHD complications, like infective endocarditis, resulting in higher morbidity/mortality. Gender disparities in VHD remains understudied, despite inequalities in risks, diagnosis, and treatment. Prevalence varies by gender, but uneven diagnostics and therapies obscure realities. This registry will examine gender disparities from hospital admission to first outpatient follow-up, recruiting both men and women to investigate and report the study objectives.

DETAILED DESCRIPTION:
Valvular heart disease (VHD) is a major global public health problem (1). Many regions of the world continue to grapple with the adverse consequences of untreated rheumatic heart disease, a condition that is largely preventable with timely access to diagnosis and treatment (2, 3). In turn, middle- and high-income countries have experienced a rise in the prevalence of calcific aortic and mitral disease, owing in part to population ageing (3). This public health problem is further compounded by high rates of infective endocarditis, which is associated with substantial morbidity and mortality. Yet, considerations of gender disparities have not taken centre stage in VHD research. This is despite evidence of major healthcare disparities in socioeconomic and medical risk factors, access to diagnosis, and provision of appropriate treatment (4-7). The prevalence of VHD varies by gender, but diagnostic evaluations are not equitable across the groups, which makes the true prevalence less clear. The delivery of evidence-based treatments for VHD is not equitable (8). The aim of this registry will be to examine gender differences in VHD from the time point of admission to the hospital (either elective or urgent admission) up to the first follow-up in an outpatient clinic. We will recruit both men and women in order to analyse the gender disparities.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diagnosis of any VHD according to the current ESC guidelines.
* Admission to the VHD-W Registry collaborating center.

Exclusion Criteria:

* Age less than 18 years old.
* Inability to provide informed consent per local institutional and regulatory requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of approximately 800 adult patients older than 18 years, with moderate-to-severe valvular heart disease (VHD) who can provide the necessary consent according to the regional/local ethical and regulatory requirements. Patients are recruited from more than 70 centers across 32 countries in Europe, America, Africa, and Australia, ensuring a diverse cohort. Eligibility includes any subtype of VHD, regardless of prior interventions, as long as the admission (urgent or elective) to a VHD-W Registry collaborating center is for management of their VHD. Collaborating Centers were invited directly by the VHD-W executive committee, supplemented by social media promotion through professional healthcare networks to encourage collaboration with centres of excellence around the globe.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Disparities in Valvular Heart Disease (VHD) Treatment | One year
  Assess disparities in evidence-based VHD treatments (medical, interventional or surgical management) by gender, in relation to age, ethnicity, and location. Quantify using odds ratios (OR) or relative risks (RR) with 95% CI; adjust via multivariable logistic regression. Time Frame: Baseline to 12 months post-enrollment. Analysis Plan: Chi-square/ANOVA for unadjusted comparisons; regression for adjusted analyses (p < 0.05).
Disparities in Valvular Heart Disease Management | One year
  Evaluate disparities in diagnostic testing, follow-up, and multidisciplinary care using composite scores and standardized mean differences (SMD) or hazard ratios (HR); adjust with Cox models if time-dependent. Time Frame: Baseline to 12 months post-enrollment. Analysis Plan: Generalized linear mixed model (GLMM) for clustering; power for Cohen's d > 0.3.
Adherence to/Compliance with European Society of Cardiology (ESC) Guidelines for Management of Valvular Heart Disease. | One Year
  Measure proportion adhering to 2021 ESC guidelines (or updates); binary/ordinal scoring with reasons for non-compliance categorized. Time Frame: Through study timepoints. Analysis Plan: Binomial proportions with 95% CI; logistic regression for predictors; detect differences.

SECONDARY OUTCOMES:
Time from Diagnosis to Guideline-Directed Therapy: Comparison Between Women and Men | One Year
  Compare median days from diagnosis to therapy initiation (medical/intervention/surgery) by sex/gender. Time Frame: Study duration. Analysis Plan: Kaplan-Meier/log-rank; Cox HR with 95% CI.
Time from Symptom Onset to Presentation at Tertiary Center: Comparison Between Women and Men | One Year
  Compare median days from symptom onset to tertiary presentation by gender. Time Frame: Study duration. Analysis Plan: Wilcoxon rank-sum; quantile regression.
Procedural Complications: Comparison Between Women and Men | One Year
  Compare reported complication post-intervention quantitatively based on established criteria or occurrence of major cardiovascular events. Time Frame: Intra/Post-procedure through study duration. Analysis Plan: Chi-square/Fisher's; Poisson IRR.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Grapsa, MD PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Ana G Almeida, MD PhD, Principal Investigator — Lisbon University
Locations (2):
- Aswan Heart Centre, Aswān, Egypt
- University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns under international regulations such as GDPR and HIPAA, which prioritize participant confidentiality in this multicenter, global registry. Data is pseudonymized for internal analysis only, and sharing could risk re-identification, especially across diverse jurisdictions with varying ethical requirements.